CLINICAL TRIAL: NCT05311267
Title: Effects of Action Observation Training (AOT) in the Achievement of Urinary Continence in Men After Robot-assisted Laparoscopic Prostatectomy (RALP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 751
Record Dates: First submitted 2022-03-11; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Urinary Incontinence
Keywords: Robot-assisted Laparoscopic Prostatectomy; Action Observation Training; pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AOT (Experimental): Participants who, in addiction to standard rehabilitation program after surgery (isometric exercises), underwent two training session of action observation therapy.
  Interventions: Other: Action observation training
- Control group (No Intervention): Participants who received standard rehabilitation program after surgery. The control group, before performing the functional exercises watched two videos of different landscapes lasting 4 minutes each.

INTERVENTIONS:
Other: Action observation training — Subject is asked to observe videos with motor contents
  Arms: AOT

SUMMARY:
Urinary incontinence (UI) is one of the most common side effects of radical prostatectomy (RP) and compromises men's quality of life. The first line treatment for urinary incontinence is the conservative approach of Pelvic Floor Muscle Training (PFMT) but, up to date, there seems to be no statistically significant difference in the effectiveness of several proposed physiotherapy treatments.

Literature highlights the importance of also adding an educational component regarding the intentional contraction of the pelvic floor muscles (a skill termed "the Knack"). Moreover, in some studies, carried out on a sample of women, was introduced the use of virtual reality. This increased the adherence to treatment and showed an improvement in urinary continence. In addition to virtual reality, another intervention methodology used in physiotherapy is the one of Action Observation training (AOT) whose effectiveness has been proven both in sports and rehabilitation.

However, currently the effect of this innovative type of treatment has not yet been studied in men with UI following radical prostatectomy intervention.

The aim of this clinical study is to investigate the effectiveness of using AOT on urinary incontinence in subjects undergoing robotic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone Robot-assisted Laparoscopic Prostatectomy with post-operative IU.
* Objectivity of recruitment and contraction of pelvic floor musculature (PP) at manual perineal testing.

Exclusion Criteria:

* Preoperative incontinence
* Pre-intervention radiotherapy
* Previous urogenital surgery beyond Robot-assisted Laparoscopic Prostatectomy.
* Concomitant presence of neurological, internal or musculoskeletal diseases that may affect functional or motor recovery.
* Less than 5 seconds of endurance in PP contraction

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 92 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Changes in continence using "24 hours pad test" | Both groups will be evaluated 45 days after surgery (T0), 1-week after T0 (T1), 2 weeks after T0 (T2), 4 weeks after T0 (T4), 6 weeks after T0 (T6) and 8 weeks after T0 (T8), 3 months after T8 (T9).
  The primary outcome is to investigate if there is a difference in continence between the experimental and the control group at each physiotherapy session and compared to the baseline (T0).To quantify the extent of these losses, the weight of absorbent devices used by patients in the 24 hours prior to each evaluation will be measured.

SECONDARY OUTCOMES:
Changes in urinary symptoms using International Prostatic Symptoms Score (IPSS) | Both groups will be evaluated 45 days after surgery (T0), 8 weeks after T0 (T8) or earlier in case of achievement of the primary goal in previous sessions (T1, T2, T4, T6), and 3 months after T8 (T9).
  The secondary objective is to investigate urinary symptoms using International Prostatic Symptoms Score (IPSS)
Changes in the quality of life using quality life index (QoL index) 0-6 | Both groups will be evaluated 45 days after surgery (T0), 8 weeks after T0 (T8) or earlier in case of achievement of the primary goal in previous sessions (T1, T2, T4, T6), and 3 months after T8 (T9).
  The secondary objective is to investigate the quality of life using quality life index 0-6
Changes in urinary symptoms using International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | Both groups will be evaluated 45 days after surgery (T0), 8 weeks after T0 (T8) or earlier in case of achievement of the primary goal in previous sessions (T1, T2, T4, T6), and 3 months after T8 (T9).
  The secondary objective is to investigate urinary symptoms using International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy